CLINICAL TRIAL: NCT06594081
Title: Use of Podcasts in Nursing Education
Acronym: PNRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Bahar Ciftci, Associate Prof, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023-3/3
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nursing Students
Keywords: nursing student

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No application will be made.
- Intervention (Experimental): Training was provided via podcast.
  Interventions: Behavioral: Intervention podcasts

INTERVENTIONS:
Behavioral: Intervention podcasts — Students in the experimental group will listen to podcasts.
  Arms: Intervention

SUMMARY:
Use of Podcasts in Nursing Education: A Randomized Controlled Trial

ELIGIBILITY:
Inclusion Criteria:

* Students who use Spotify
* Those who have a smart phone
* Those who have enough internet connection to listen to podcasts on Spotify
* Students taking the Fundamentals of Nursing course for the first time
* Students who are not horizontal/vertical transfer students
* Students who have not graduated from Health Vocational High School
* Those who were not absent during the study were included in the study.

Exclusion Criteria:

* Students who were not first-year nursing students
* Students who did not use Spotify
* Students who came via horizontal/vertical transfer
* Students who graduated from Health Vocational High School
* Students in the intervention group who did not listen to podcasts on Spotify
* Students in the control group who were understood to have logged into their Spotify accounts and listened to podcasts were excluded from the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Motivation Scale Related to Instructional Material | 6 months
  "ÖMMÖ" is a 33-item four-dimensional (attention, suitability, trust, satisfaction) measurement tool that evaluates the entire course in order to measure motivation towards the teaching material, developed by Keller based on the ARCS (Attention, Relevance, Confidence, Satisfaction) Model, and adapted into Turkish by Dinçer and Doğanay. The original scale contains 36 items. The scale was prepared in a 5-point Likert type and is scored as "Very True" 5, "True" 4, "Moderately True" 3, "Somewhat True" 2, and "Not True" 1. The highest score that can be obtained from the entire scale is 165, and the lowest score is 33. The highest score that can be obtained from the attention dimension is 50, and the lowest score is 10. The highest score that can be obtained from the suitability dimension is 40, and the lowest score is 8. The highest score that can be obtained from the confidence dimension is 45, and the lowest score is 9. The highest score that can be obtained from the satisfaction dimensio

SECONDARY OUTCOMES:
"Achievement Test 1" and "Achievement Test 2" | 6 months
  Multiple choice questions were prepared by the researchers after a literature review. The questions in "Achievement Test 1" and "Achievement Test 2" related to the subject of "Parenteral drug applications" were created in a way that they would be different from each other. After the questions were created, expert opinions were received from a total of 10 faculty members working in the nursing fundamentals department (7) and nursing education department (3). After the necessary suggestions for the questions presented to the experts were arranged, the achievement tests were finalized. 25 of the 50 multiple choice questions were duplicated as many times as the number of students for "Achievement Test 1" and "Achievement Test 2" and kept ready before the application. "Achievement Test 1" was applied to the students who would participate in the study by taking them to separate classes. The evaluation of the achievement tests was made out of 100 points. For this purpose, the students' total

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Çiftçi, Study Director — Ataturk University
Locations (1):
- Bahar Çiftçi, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No